CLINICAL TRIAL: NCT02580851
Title: Magnetic Resonance Adenosine Perfusion Imaging as Gatekeeper of Invasive Coronary Intervention
Acronym: MAGnet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Dr. Dominik Buckert, MD, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 237/11
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Stable Coronary Artery Disease; Cardiac Magnetic Resonance Imaging; Coronary Angiography; Myocardial Revascularization; Outcomes and Prognosis; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coronary angiography (Other): Patients directly undergo diagnostic coronary angiography. A PCI is performed according to current guidelines in case of ≥70% stenosis in a coronary vessel with ≥2 mm diameter.
  Interventions: Other: diagnostic test - coronary angiography
- Cardiac magnetic resonance imaging (Other): Patients receive adenosine perfusion CMR for functional testing, first. The examination is conducted on a 3.0 Tesla whole-body scanner with a 32-channel phased-array cardiac receiver coil according to a well-established standard protocol [21-23]. In case reversible ischemia can be detected, subjects are sent to coronary angiography and PCI afterwards.
  Interventions: Other: diagnostic test - cardiac magnetic resonance imaging

INTERVENTIONS:
Other: diagnostic test - cardiac magnetic resonance imaging
  Arms: Cardiac magnetic resonance imaging
Other: diagnostic test - coronary angiography
  Arms: Coronary angiography

SUMMARY:
Current guidelines for the diagnosis and management of patients with stable coronary artery disease (CAD) strongly support the performance of non-invasive imaging techniques for the detection of myocardial ischemia prior to revascularization procedures. This recommendation originates from the strong evidence base showing the lack of prognostic benefit from percutaneous coronary interventions (PCI) over optimal medical therapy in patients without verification of myocardial ischemia. On the other hand, it could be demonstrated that patients with functionally significant coronary artery stenoses do benefit from revascularization. Cardiac magnetic resonance imaging (CMR) has emerged to be a diagnostic modality of choice for the detection of myocardial ischemia with high sensitivity and specificity. The investigators therefore designed this prospective and randomized trial to compare a CMR-driven vs. angiography-driven management of patients with stable CAD concerning major cardiac endpoints, futile angiographies and quality of life.

DETAILED DESCRIPTION:
Current guidelines for the diagnosis and management of patients with stable coronary artery disease (CAD) recommend - besides thorough history and physical examination - proper risk stratification prior to invasive therapy. The detection or exclusion of moderate to severe reversible myocardial ischemia is a crucial part of the work-up process which designates the patients to the high-risk group when ischemia is present. This is of special interest, as several observational studies have shown that the prognostic benefit from revascularization depends on the amount of myocardial ischemia. Moreover, patients without ischemia do not seem to benefit from revascularization over optimal medical therapy. This emphasizes the need for functional testing prior to therapeutic decisions.

Invasive coronary angiography still is considered to be the "gold-standard" for the diagnosis of CAD, though it exhibits several limitations and shortcomings. Multiple studies have documented the significant interobserver variability in the grading of coronary artery stenosis, as well as the frequent occurrence of under- and overestimation of hemodynamic relevance. One has to conclude that coronary angiography may provide anatomical information but is not the modality of choice concerning the detection of myocardial ischemia. Moreover, there is no study which has randomized patients with stable CAD to either catheterization or no catheterization yet, so there does not exist high-quality evidence which would support the performance of a diagnostic coronary angiography in the majority of cases of stable CAD. This is of special interest, as there is a reported frequency of complications due to diagnostic coronary angiography of about 1.5%. Nevertheless, coronary angiography remains the most often performed diagnostic test in this setting, with more than one-half of elective percutaneous coronary interventions (PCI) done without previous stress-testing.

Adenosine perfusion cardiac magnetic resonance imaging (CMR) is an imaging modality which provides anatomical and functional information in one single examination. With its ability to reliably detect reversible myocardial ischemia, it plays an increasing role in the diagnosis and risk stratification of patients with suspected or known CAD. Though CMR therefore is highly recommended in the diagnostic work-up in the setting of stable CAD, no study exists which would have evaluated a CMR driven approach in patient management with regard to the occurrence of major cardiac events, quality of life and safety endpoints.

Objective of our study is to show that a CMR based conservative or invasive management of patients with suspected or known CAD is not inferior with regard to major cardiac endpoints and quality of life in comparison to a - more conventional - coronary angiography based approach. The investigators assume that a significant number of diagnostic coronary angiographies and PCIs thus could be spared without decrease in patient safety and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present themselves for the evaluation of symptoms being likely to be caused by CAD, such as exercise-related chest pain or dyspnea.

Exclusion Criteria:

* Unability to give written informed consent
* Unstable angina
* Cardiac or respiratory instability
* Contraindication for CMR
* Allergy to Gadolinium
* Impaired renal function
* Allergy to adenosine
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-12; Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of cardiac deaths and non-fatal myocardial infarctions occurring in study cohort assessed by medical records | 3 years

SECONDARY OUTCOMES:
Number of invasive procedures | 3 years
  Diagnostic coronary angiographies/PCIs
Quality of life | 3 years
  Assessed by Seattle Angina Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bernhardt, Prof. Dr., Principal Investigator — University of Ulm
Locations (1):
- University of Ulm, Ulm, Germany

REFERENCES:
- [Derived] Buckert D, Witzel S, Steinacker JM, Rottbauer W, Bernhardt P. Comparing Cardiac Magnetic Resonance-Guided Versus Angiography-Guided Treatment of Patients With Stable Coronary Artery Disease: Results From a Prospective Randomized Controlled Trial. JACC Cardiovasc Imaging. 2018 Jul;11(7):987-996. doi: 10.1016/j.jcmg.2018.05.007. PMID 29976305
- [Derived] Buckert D, Witzel S, Cieslik M, Tibi R, Rottbauer W, Bernhardt P. Magnetic resonance Adenosine perfusion imaging as Gatekeeper of invasive coronary intervention (MAGnet): study protocol for a randomized controlled trial. Trials. 2017 Jul 28;18(1):358. doi: 10.1186/s13063-017-2101-6. PMID 28754155